CLINICAL TRIAL: NCT03486938
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of AGB101on Slowing Progression of Mild Cognitive Impairment Due to Alzheimer's Disease
Brief Title: Study of AGB101 in Mild Cognitive Impairment Due to Alzheimer's Disease
Acronym: HOPE4MCI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AgeneBio (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AGB101 MCD; R56AG055416 (NIH); R01AG048349 (NIH); R01AG061091 (NIH)
Record Dates: First submitted 2018-03-28; First posted 2018-04-03 (Actual); Results first posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Mild Cognitive Impairment; Prodromal Alzheimer's Disease
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo Oral Tablet (Placebo Comparator): Matching placebo to AGB101 tablet once daily, taken orally, for 78 weeks.
  Interventions: Drug: Placebo Oral Tablet
- AGB101 220 mg tablet (Experimental): Single 220 mg AGB101 tablet once daily, taken orally, for 78 weeks.
  Interventions: Drug: AGB101 220 mg tablet

INTERVENTIONS:
Drug: Placebo Oral Tablet — Placebo oral tablet
  Arms: Placebo Oral Tablet
Drug: AGB101 220 mg tablet — 220 mg AGB101 active compound
  Arms: AGB101 220 mg tablet

SUMMARY:
The primary objective of the study is to evaluate the efficacy of AGB101 on slowing cognitive and functional impairment as measured by changes in the Clinical Dementia Rating-Sum of Boxes (CDR-SB) score as compared with placebo in participants with mild cognitive impairment due to Alzheimer's Disease (MCI due to AD) also known as prodromal AD. Participants will be randomized to receive placebo or AGB101 (220 mg), once daily for 78 weeks. Secondary objectives are to assess the effect of AGB101 compared with placebo on clinical progression as measured by Mini-Mental State Examination (MMSE) and Functional Activities Questionnaire (FAQ).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects between 55 and 85 years old (inclusive) in good general health:

   1. Willing and able to consent and participate for the duration of the study
   2. Have eighth-grade education or good work history sufficient to exclude mental retardation
   3. Have visual and auditory acuity adequate for neuropsychological testing
   4. Have proficient fluency of the native local language to participate in all the neuropsychological test assessments
2. Have a study partner who has sufficient contact with the subject to be able to provide assessment of memory changes, who can accompany the subject to all the clinic visits for the duration of each visit, and who is able to provide an independent evaluation of the subject's functioning
3. Have MCI due to AD as defined by all of the following criteria and consistent with the National Institute on Aging-Alzheimer's Association criteria:

   1. MMSE scores between 24 and 30 (inclusive; exceptions may be made for subjects with <8 years of education at the discretion of the sponsor)
   2. A memory complaint reported by the subject or his/her study partner
   3. Evidence of lower memory performance based on delayed recall in the International Shopping List Test (ISLT)
   4. A clinical dementia rating (CDR) score of 0.5 with a memory box score of ≥0.5
   5. Essentially preserved activities of daily living
   6. Cognitive decline not primarily caused by vascular, traumatic, or medical problems (alternative causes of cognitive decline are ruled out)
4. Permitted medications:

   1. With potential pro-cognitive effects, such as cholinesterase inhibitors and memantine, must be at a stable dose for ≥3 months prior to screening and remain stable throughout the study; estrogen replacement therapy, Ginkgo biloba, and vitamin E must be at a stable dose for ≥4 weeks prior to screening and remain stable throughout the study
   2. Other psychotropics, such as antidepressants and antipsychotics, must be at a stable dose for ≥3 months prior to screening and remain stable throughout the study
5. Willing and able to undergo imaging procedures:

   1. A Positron Emission Tomography (PET) scan with Florbetaben(an 18F isotope diagnostic agent) or documented evidence of an amyloid positive PET scan.

      The Florbetaben scan performed at baseline must be read by a qualified physician with experience in reading amyloid PET scans, and it should be consistent with the presence of amyloid plaques.
   2. Repeated MRI scans (3 Tesla) with no contraindications to MRI. MRI scan results are consistent with the diagnosis of amnestic MCI due to Alzheimer's disease with no clinically significant findings of non-AD pathology that could account for the observed cognitive impairment.
6. Willing to allow collection of blood for apolipoprotein E (ApoE) genotyping.

Exclusion Criteria:

1. Use of anticonvulsant medications or excluded psychotropic medications within 3 months prior to the baseline visit
2. Participation in a therapeutic clinical study for any medical or psychiatric indications within 3 months (6 months for biologics) of the screening visit, or at any time during the study.

   Subjects must understand that they may only enroll in this clinical study once; they may not enroll in any other clinical study while participating in the current study, and they may not participate in a clinical study of a drug, biologic, therapeutic device, or medical food, in which the last dose/administration was received within 3 months (6 months for biologics) prior to screening.
3. History of hypersensitivity or lack of tolerability to AGB101 (levetiracetam)
4. Severe renal impairment (creatinine clearance of <30 mL/minute) or undergoing hemodialysis
5. Any significant neurological disease other than suspected incipient AD, such as Parkinson's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder (lifetime history; infant febrile seizures are not exclusionary), subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic deficits, or known structural brain abnormalities
6. Presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments, or foreign objects in the eyes, skin, or body
7. Diagnosis of major depression or bipolar disorder, as described in the Diagnostic and Statistical Manual of Mental Disorders, 5th Ed (DSM-5), within the past 3 years.

   Psychotic features, agitation, or behavioral problems within the last 3 months that could lead to difficulty complying with the protocol. Subjects must not have a major depressive disorder or other types of depression that could confound diagnosis of MCI due to AD, or clinical assessments, in the opinion of the investigator. The geriatric depression scale (long form score >9 suggests depression) results should be reviewed by the investigator to assist in this determination.
8. Modified Hachinski Ischemic Scale (HIS) score >4
9. History of schizophrenia (DSM-5 criteria)
10. History of alcohol or substance abuse or dependence within the past 3 years (DSM-5 criteria)
11. Any significant systemic illness or unstable medical condition that could lead to difficulty in complying with the protocol requirements.
12. Clinically significant abnormalities in B12 or thyroid function test that might interfere with the study.

    A low B12 (below normative range for elderly) is exclusionary, unless follow-up labs (homocysteine and methylmalonic acid) indicate that it is not physiologically significant. If the B12 deficiency is treated, subjects may become eligible to participate in the study.
13. Residence in a skilled nursing facility. Individuals in independent living communities, assisted living facilities, residential care facilities, or continuing care communities are eligible provided they engage in a sufficient spectrum of activity to permit assessment of all 6 domains contributing to the CDR-SB. Individuals in these facilities must also have a caregiver who has the ability to observe the subject during the study and can participate in clinical evaluations.
14. Any use of excluded medications (e.g., antiepileptics, certain antidepressants or antipsychotics, antihistamines with anticholinergic properties, opiates)
15. Participation in clinical studies using the ISLT, Behavioral Pattern Separation (BPS-O) task, or the trail making test (A, B) within 1 month of screening
16. Female subjects must not be pregnant, lactating, or of childbearing potential (i.e., they must be 2 years post menopause or surgically sterile)

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Mohs, PhD, Principal Investigator — AgeneBio; Sharon Rosenzweig-Lipson, PhD, Study Director — AgeneBio; Russell Barton, MS, Study Director — AgeneBio
Locations (24):
- United States (23):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Senior Clinical Trials, Inc., Laguna Hills, California
  - Excell Research Inc, Oceanside, California
  - The Mile High Research Center, Denver, Colorado
  - Boynton Beach Medical Research Institite, Boynton Beach, Florida
  - Brain Matters Research, Delray Beach, Florida
  - MD Clinical, Hallandale, Florida
  - Miami Jewish Health, Miami, Florida
  - Bioclinica Research, Orlando, Florida
  - IMIC Research, Palmetto Bay, Florida
  - The Roskamp Institute, Inc, Sarasota, Florida
  - Brain Matters Research, Stuart, Florida
  - NeuroStudies.net, LLC, Decatur, Georgia
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Memory Center/Hattiesburg Clinic, Hattiesburg, Mississippi
  - Clinical Research Professionals, Chesterfield, Missouri
  - The NeuroCognitive Institute, Mount Arlington, New Jersey
  - Global Medical Institutes LLC; Princeton Medical Institute, Princeton, New Jersey
  - Neurology Specialist of Monmouth County, PA, West Long Branch, New Jersey
  - Neurological Associates of Albany PC, Albany, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Clinical Biotechnology Research Institute at RSFH, Charleston, South Carolina
- Toronto Memory Program, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo Oral Tablet | AGB101 220 mg Tablet
Started | 83 | 81
Completed | 66 | 55
Not Completed | 17 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Oral Tablet | AGB101 220 mg Tablet | Total
Number analyzed (Participants) | 83 | 81 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.1 (7) | 72.2 (6.7) | 72.7 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 32 | 72
  Male | 43 | 49 | 92
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 81 | 75 | 156
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Clinical Dementia Rating-Sum of Boxes (CDR-SB) [Mean (Standard Deviation); unit: units on a scale] — The CDR-SB is the sum score of 6 domains of cognitive function (memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care), with the score of each domain ranging from 0 (no impairment) to 3 (severe impairment). The total possible range is 0 to 18 with higher scores indicating greater impairment.
  units on a scale | 2.7 (1.1) | 2.7 (1) | 2.7 (1)
Mini Mental Status Exam (MMSE) [Mean (Standard Deviation); unit: units on a scale] — The MMSE is the sum score of an 11 item exam designed to assess five components of cognition: orientation, registration, attention and calculation, recall, and language. The total possible range is 0-30, with lower scores indicating greater impairment.
  units on a scale | 26 (2.2) | 26.2 (2.1) | 26.1 (2.1)
Functional Activities Questionnaire (FAQ) [Mean (Standard Deviation); unit: units on a scale] — The FAQ measures instrumental activities of daily living, such as preparing balanced meals and managing finances. The total possible range is from 0 to 30, with higher scores indicating greater impairment. Population: Baseline FAQ measure not collected for 7 subjects.
  units on a scale
    number analyzed (Participants) | 81 | 76 | 157
    (all) | 7.0 (5.2) | 7.6 (5.5) | 7.3 (5.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinical Dementia Rating Scale - Sum of Boxes (CDR-SB) Score From Baseline
Description: CDR-SB scores at baseline were subtracted from CDR-SB scores at week 78 to generate the change score from baseline, with a possible total range of -18 to 18. Positive change scores reflect greater impairment on the CDR-SB at week 78, while negative change scores reflect less impairment on the CDR-SB at week 78.
Time Frame: 78 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Oral Tablet | AGB101 220 mg Tablet
Number analyzed (Participants) | 83 | 81
score on a scale | 1.1 (2) | .9 (1.5)

2. Secondary Outcome: Change in Mini Mental Status Exam (MMSE) Score From Baseline
Description: MMSE scores at baseline were subtracted from MMSE scores at week 78 to generate the change score from baseline, with a possible total range of -30 to 30. Positive change scores reflect improved performance on the MMSE at week 78, while negative change scores reflect worsening performance on the MMSE at week 78.
Time Frame: 78 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Oral Tablet | AGB101 220 mg Tablet
Number analyzed (Participants) | 83 | 81
units on a scale | -1.9 (3.7) | -2.2 (2.8)

3. Secondary Outcome: Change in Functional Activities Questionnaire (FAQ) Score From Baseline
Description: FAQ scores at baseline were subtracted from FAQ scores at week 78 to generate the change score from baseline, with a possible total range of -30 to 30. Positive change scores reflect greater impairment on the FAQ at week 78, while negative change scores reflect less impairment on the FAQ at week 78.
Time Frame: 78 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Oral Tablet | AGB101 220 mg Tablet
Number analyzed (Participants) | 83 | 81
units on a scale | 3.6 (6.4) | 4 (5.3)

ADVERSE EVENTS:
Time Frame: 18 months
Description: Three subjects were randomized and assigned to receive AGB101 but were not treated, lowering the total number of at risk participants treated with AGB101 to 78.
Arm/Group | Placebo Oral Tablet | AGB101 220 mg Tablet
All-Cause Mortality (participants affected / at risk) | 0/83 | 2/78
Serious Adverse Events (participants affected / at risk) | 10/83 | 13/78
Other Adverse Events (participants affected / at risk) | 49/83 | 40/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Oral Tablet (N=83) | AGB101 220 mg Tablet (N=78)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 3 (3)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia legionella (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 2 (2)
Transient ischemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive urgency (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Oral Tablet (N=83) | AGB101 220 mg Tablet (N=78)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 7 (8) | 2 (2)
cardiac disorders (Cardiac disorders) | 3 (7) | 1 (5)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Endocrine disorders (Endocrine disorders) | 0 (0) | 1 (1)
Eye disorders (Eye disorders) | 3 (3) | 1 (2)
Gastrointestinal disorders (Gastrointestinal disorders) | 13 (18) | 7 (10)
General disorders and administration site condition (General disorders) | 10 (14) | 5 (5)
Hepatobiliary disorders (Hepatobiliary disorders) | 1 (1) | 1 (1)
Infections and infestations (Infections and infestations) | 13 (19) | 11 (12)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 15 (31) | 12 (18)
Investigations (Investigations) | 8 (8) | 7 (7)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 6 (7) | 5 (7)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 20 (31) | 11 (14)
Neoplasms benign, malignant and unspecified (inc cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (9) | 2 (2)
Nervous system disorders (Nervous system disorders) | 15 (21) | 8 (15)
Product issues (Product Issues) | 0 (0) | 1 (1)
Psychiatric disorders (Psychiatric disorders) | 9 (11) | 14 (21)
Renal and urinary disorders (Renal and urinary disorders) | 2 (5) | 1 (1)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 2 (2)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 7 (7) | 2 (2)
Social circumstances (Social circumstances) | 1 (1) | 0 (0)
Surgical and medical procedures (Surgical and medical procedures) | 1 (2) | 1 (1)
Vascular disorders (Vascular disorders) | 7 (7) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-19): https://cdn.clinicaltrials.gov/large-docs/38/NCT03486938/Prot_SAP_000.pdf